CLINICAL TRIAL: NCT05314569
Title: Cardioprotective Effect of Ketamine-dexmeditomidine Versus Fentanyl-midazolam in Open-heart Surgery in Pediatrics: A Randomized Controlled Double-blinded Study
Brief Title: Cardioprotective Effect of Ketamine-dexmeditomidine Versus Fentanyl-midazolam in Open Heart Surgery in Pediatrics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Associate professor of anesthesia ,surgical intensive care and pain management ,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N-11-2022
Record Dates: First submitted 2022-03-27; First posted 2022-04-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Isoflurane

STUDY DESIGN:
Intervention Model Description: patients will be allocated to three groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: patients will be allocated to the study using a computer-generated random list and the group assignments will be sealed in opaque envelopes that will be opened after induction. The drugs will be prepared by an anesthetist who is blind to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group(C) (Placebo Comparator): anesthesia will be maintained using Isoflurane 1.2MAC keeping the bispectral index( BIS) between 40-60%.
  Interventions: Drug: Isoflurane
- Ketamine-dexmedetomidine group( KD) (Active Comparator): After induction of anesthesia , dexmedetomidine will be given(1 ug /kg ) over 10 min, then ketamine(2 m/kg) . maintenance throughout the procedure, with the bispectral index between 40 and 60%. by infusing Dexmedetomidine( 0.5 μg/.kg /.h r)) ketamine,( 1 m/kg/hr),
  Interventions: Drug: Ketamine- dexmedetomidine
- . Fentanyl- midazolam group (FM) (Active Comparator): After induction of anesthesia fentanyl( 3 μg/kg), midazolam( 100 ug /kg over 2 to 3 minutes) maintenance throughout the procedure, with the bispectral index between 40 and 60%. by infusing midazolam (1 ug /kg /min)-fentanyl( 2 μg/kg/h ).
  Interventions: Drug: Fentanyl- midazolam

INTERVENTIONS:
Drug: Ketamine- dexmedetomidine — ketamine - Dexmedetomidine combination had superior cardioprotective effects as measured by cardiac markers as compared to sevoflurane- sufentanil anesthesia after cardiac surgery
  Arms: Ketamine-dexmedetomidine group( KD)
Drug: Fentanyl- midazolam — Midazolam is known to have potential anti-inflammatory effects and antioxidant activity. They have been proven to provide protective effects for patients who underwent cardiac surgery.Fentanyl is one opioid that has been closely linked to inflammatory mediators and myocardial protection. It reduces the CPB-induced inflammatory response and ischaemic reperfusion injury during cardiac surgery
  Arms: . Fentanyl- midazolam group (FM)
Drug: Isoflurane — Anesthetic inhalational gas
  Arms: Control group(C)

SUMMARY:
congenital hearts are very sensitive and irritable to deal with, especially during repair defects, the child's heart is exposed to impaired myocardial function during the entire procedure. Moreover, reperfusion of the heart during open-heart surgery when the myocardium is exposed to a global ischaemic cardioplegic arrest can induce myocardial injury. Myocardial reperfusion injury activates neutrophils, which trigger an inflammatory response resulting in the generation of reactive oxygen species (ROS), cytokine release, and complement activation, which further induce more cardiac injury. In addition to the inflammatory response generated as a result of tissue reperfusion injury, there is a significant systemic inflammatory response that is triggered by cardiopulmonary bypass (CPB) during open-heart surgery

DETAILED DESCRIPTION:
Myocardial protection is an important issue. This is reflected in the clinical prognosis of patients undergoing cardiac surgery and this can be measured by the most popular Cardiac biomarkers ( cardiac troponin I (cTnI)). (2)

A large number of anesthetic agents have been implicated in protecting the heart against ischemia and reperfusion injury. Ketamine has an anti-inflammatory effect and has been shown to reduce ROS generation by neutrophils and to decrease endotoxin stimulated IL6 production in human whole blood although it does not impair neutrophil function. (3)

Dexmedetomidine is a highly selective, short-acting, central α2-adrenergic agonist with intense sympatholytic qualities. Dexmedetomidine has been increasingly used as a component of general anesthesia, including cardiac surgical applications due to its sedative/hypnotic and analgesic effects which are enhanced by its cardioprotective properties. (4) Riha et.al showed that ketamine - Dexmedetomidine combination had superior cardioprotective effects as measured by cardiac markers as compared to sevoflurane- sufentanil anesthesia after cardiac surgery. (5) Midazolam is known to have potential anti-inflammatory effects and antioxidant activity. They have been proven to provide protective effects for patients who underwent cardiac surgery. (6) Fentanyl is one opioid that has been closely linked to inflammatory mediators and myocardial protection. It reduces the CPB-induced inflammatory response and ischaemic reperfusion injury during cardiac surgery. These effects are related to improvement in intracellular Ca2+ mobilization and do not seem to be related to the adhesion of neutrophils in the coronary system. (7) To the best of our knowledge, this is the first study comparing the combined effect of Ketamine- Dexmedetomidine versus fentanyl- midazolam against ischemia and reperfusion injury in pediatric congenital heart surgery repair.

ELIGIBILITY:
Inclusion Criteria:

* the American Society of Anesthesiologists II and III
* elective open Congenital cardiac surgery(VSD, AV canal, and partial anomaly) using cardiopulmonary bypass

Exclusion Criteria:

* less than 6 months or more than 24 months.
* weight < 5 kg.
* cyanotic heart disease
* patients with heart failure, an implantable pacemaker, pulmonary hypertension, preoperative administration of inotropic agents, serum creatinine higher than1.5 mg/dL, chronic liver disease, patients receiving sulfonylurea, theophylline, or allopurinol

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
troponin level | 6 hours
  mean troponin level post arotic declamping.

SECONDARY OUTCOMES:
heart rates | every 15 minutes
  records of reading till the end of the surgery
aortic cross clamping | 2 hours
  duration of clamping
inotropic support | 6 hours
  number of patients
blood pressure | every 15 minutes
  records of reading till the end of the surgery
need of nitroglycerin infusion | 6 hours
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Amany H Saleh, MD, Principal Investigator — Cairo University
Locations (1):
- Amany Hassan Saleh, Giza, Egypt